CLINICAL TRIAL: NCT00312117
Title: A Randomized Trial for Prevention of Contrast Nephropathy With Sodium Bicarbonate
Brief Title: Trial for Prevention of Contrast Nephropathy With Sodium Bicarbonate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 4353
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Contrast Induced Nephropathy; Kidney Diseases
Keywords: contrast induced nephropathy; sodium bicarbonate; cardiac catheterization
MeSH Terms: conditions — Kidney Diseases | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sodium bicarbonate

SUMMARY:
Contrast nephropathy (CN) is a common cause of renal failure associated with prolonged hospitalization, significant morbidity/mortality, and cost. In addition, these patients may require temporary or permanent hemodialysis which, in turn, is associated with further morbidity, mortality, and cost. CN has been reported to account for 10% of hospital acquired renal failure. In recent years, studies have investigated preventive therapies with mixed results. Fenoldopam was found to be ineffective in a large randomized trial. Dopamine has been shown to be ineffective as a preventive strategy. Hemofiltration has been shown to be beneficial (New England Journal of Medicine [NEJM] 2003) but is costly and not practical. Mucomyst has shown mixed results. The single strategy which most would agree as being beneficial remains hydration, most commonly with intravenous 0.9% normal saline. Most recently, sodium bicarbonate has been shown to be beneficial in a small randomized trial (n=119). It is clear that the most cost effective strategies for treatment of CN should be aimed at prevention.

The general question is: "Is a sodium bicarbonate solution more efficacious in preventing contrast nephropathy compared to normal saline?" The general hypothesis is that sodium bicarbonate will be more efficacious.

ELIGIBILITY:
Inclusion Criteria:

* GFR < 60 mL/min/1.73m2. GFR will be adjusted by a correction factor as reported by our laboratory for patients self identifying as black.
* > 18 years and have at least one of the following risk factors for contrast nephropathy: diabetes (type 2), congestive heart failure, hypertension (> 140/90), or age > 75.
* Both inpatients and outpatients will be offered enrollment.

Exclusion Criteria:

* Patients unable to give consent
* Already receiving sodium bicarbonate solution
* Undergoing emergency cardiac catheterization
* Receiving a contrast agent other than Oxilan
* On hemodialysis
* Recent exposure to contrast within 2 days
* Pulmonary edema
* Active congestive heart failure
* Severe valvular abnormality
* Recent significant change in kidney function (> 15% over 2d)
* One kidney
* Kidney transplant status

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2006-01; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
development of contrast induced nephropathy, defined by a decrease in glomerular filtration rate (GFR) by 25% or more

SECONDARY OUTCOMES:
change in serum creatinine
difference in hospital duration between groups
need for hemodialysis
30 day mortality
difference of baseline to lowest GFR and highest creatinine between groups
difference in GFR and creatinine from baseline and 2-8 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Somjot S Brar, M.D., Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Briguori C, Tavano D, Colombo A. Contrast agent--associated nephrotoxicity. Prog Cardiovasc Dis. 2003 May-Jun;45(6):493-503. doi: 10.1053/pcad.2003.YPCAD16. PMID 12800130
- [Background] McCullough PA, Wolyn R, Rocher LL, Levin RN, O'Neill WW. Acute renal failure after coronary intervention: incidence, risk factors, and relationship to mortality. Am J Med. 1997 Nov;103(5):368-75. doi: 10.1016/s0002-9343(97)00150-2. PMID 9375704
- [Background] Marenzi G, Lauri G, Assanelli E, Campodonico J, De Metrio M, Marana I, Grazi M, Veglia F, Bartorelli AL. Contrast-induced nephropathy in patients undergoing primary angioplasty for acute myocardial infarction. J Am Coll Cardiol. 2004 Nov 2;44(9):1780-5. doi: 10.1016/j.jacc.2004.07.043. PMID 15519007
- [Background] Merten GJ, Burgess WP, Gray LV, Holleman JH, Roush TS, Kowalchuk GJ, Bersin RM, Van Moore A, Simonton CA 3rd, Rittase RA, Norton HJ, Kennedy TP. Prevention of contrast-induced nephropathy with sodium bicarbonate: a randomized controlled trial. JAMA. 2004 May 19;291(19):2328-34. doi: 10.1001/jama.291.19.2328. PMID 15150204
- [Background] Rihal CS, Textor SC, Grill DE, Berger PB, Ting HH, Best PJ, Singh M, Bell MR, Barsness GW, Mathew V, Garratt KN, Holmes DR Jr. Incidence and prognostic importance of acute renal failure after percutaneous coronary intervention. Circulation. 2002 May 14;105(19):2259-64. doi: 10.1161/01.cir.0000016043.87291.33. PMID 12010907
- [Background] Parfrey PS, Griffiths SM, Barrett BJ, Paul MD, Genge M, Withers J, Farid N, McManamon PJ. Contrast material-induced renal failure in patients with diabetes mellitus, renal insufficiency, or both. A prospective controlled study. N Engl J Med. 1989 Jan 19;320(3):143-9. doi: 10.1056/NEJM198901193200303. PMID 2643041
- [Derived] Brar SS, Shen AY, Jorgensen MB, Kotlewski A, Aharonian VJ, Desai N, Ree M, Shah AI, Burchette RJ. Sodium bicarbonate vs sodium chloride for the prevention of contrast medium-induced nephropathy in patients undergoing coronary angiography: a randomized trial. JAMA. 2008 Sep 3;300(9):1038-46. doi: 10.1001/jama.300.9.1038. PMID 18768415